CLINICAL TRIAL: NCT00477230
Title: Pivotal Clinical Study of the CardioFocus Endoscopic Ablation System for the Treatment of Symptomatic Atrial Fibrillation (AF)
Brief Title: Pivotal Clinical Study of Endoscopic Ablation for Atrial Fibrillation (AF) in Patients That Have Failed Drugs
Acronym: ENABLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated based on decision of Sponsor.
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENABLE 25-2064
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
Keywords: AF; PAF; paroxysmal atrial fibrillation; ablation; failed drugs
MeSH Terms: conditions — Atrial Fibrillation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Single ablation procedure with Endoscopic Ablation System
  Interventions: Device: Endoscopic Ablation System
- 2 (Active Comparator): Medication
  Interventions: Drug: Standard Anti-arrhythmic Drug (AAD) Therapy

INTERVENTIONS:
Device: Endoscopic Ablation System — Single ablation procedure with Endoscopic Ablation System
  Arms: 1
Drug: Standard Anti-arrhythmic Drug (AAD) Therapy — Medication as prescribed by physician.
  Arms: 2

SUMMARY:
The purpose of the study is to compare two types of treatment for atrial fibrillation (AF) that are designed to treat the symptoms of atrial fibrillation. The treatments being compared are:

* A single catheter ablation procedure with the investigational EAS, a visually-guided, light-energy catheter
* Standard drug therapy (antiarrhythmic drugs)

To learn more about the CardioFocus ENABLE investigational clinical study, please contact the study site closest to you.

Eligibility Criteria

Persons with paroxysmal atrial fibrillation may be eligible for this study. Other study eligibility criteria include:

* 18 to 80 years of age
* Frequent episodes of AF
* Failed at least 1 drug treatment for AF (beta-blockers or standard AADs)
* Other criteria

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* Paroxysmal atrial fibrillation (AF)
* Frequent episodes of AF
* Failed at least 1 drug treatment
* Others

Exclusion Criteria:

* Others

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — University of Miami; Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia; Burke Barrett, Study Director — CardioFocus, Inc.
Locations (18):
- United States (18):
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Mercy General Hospital, Sacramento, California
  - University of California at San Francisco, San Francisco, California
  - St. John's Health Center, Santa Monica, California
  - Palm Beach Heart Research Institute, Atlantis, Florida
  - Florida Hospital, Orlando, Florida
  - Indiana University, Krannert Institute of Cardiology, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Luke's-Roosevelt, New York, New York
  - Strong Memorial Hosptial - University of Rochester, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early by the decision of the Sponsor after 64 participants were enrolled and 25 were treated.
Pre-assignment Details: None outside of the protocol.
Groups:
- Single Ablation Procedure With Endoscopic Ablation System: Single ablation procedure with Endoscopic Ablation System
- Standard Anti-arrhythmic Drug Therapy: Medication as prescribed by physician.
Period: Overall Study
Arm/Group | Single Ablation Procedure With Endoscopic Ablation System | Standard Anti-arrhythmic Drug Therapy
Started | 32 | 32
Completed | 12 | 1
Not Completed | 20 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Ablation Procedure With Endoscopic Ablation System | Standard Anti-arrhythmic Drug Therapy | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Customized [Number; unit: Participants]
  Less than 18 Years | 0 | 0 | 0
  Greater than or equal to 18 Years | 32 | 32 | 64
Sex/Gender, Customized [Number; unit: Participants]
  Male | 0 | 0 | 0
  Female | 0 | 0 | 0
  Unknown | 32 | 32 | 64
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Freedom for Symptomatic Episode of Atrial Fibrillation at One Year
Time Frame: One Year
Population: Early study termination before one year.
Measure: Number; unit: participants
Arm/Group | Single Ablation Procedure With Endoscopic Ablation System | Standard Anti-arrhythmic Drug Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: After treatment and during up to 1 year follow-up.
Arm/Group | Single Ablation Procedure With Endoscopic Ablation System | Standard Anti-arrhythmic Drug Therapy
Serious Adverse Events (participants affected / at risk) | 5/32 | 0/32
Other Adverse Events (participants affected / at risk) | 4/32 | 5/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Ablation Procedure With Endoscopic Ablation System (N=32) | Standard Anti-arrhythmic Drug Therapy (N=32)
Mechanical Perforation (Cardiac disorders) | 4 | 0
Pericarditis (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Ablation Procedure With Endoscopic Ablation System (N=32) | Standard Anti-arrhythmic Drug Therapy (N=32)
diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
chest pain (Ear and labyrinth disorders) | 2 | 0
Medication Intolerance (Injury, poisoning and procedural complications) | 0 | 5

LIMITATIONS AND CAVEATS:
This study was terminated early due to Sponsor decision. Therefore, full patient assignement to treatments post-randomziation did not occur. Results and other measures cannot be determined because most patients exited the study before completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No